CLINICAL TRIAL: NCT05575908
Title: Expert@Work - Effectiveness of a Digital Expert Team on Return to Work
Acronym: Expert@Work
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian Labour and Welfare Administration (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/11991
Record Dates: First submitted 2022-09-21; First posted 2022-10-12 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Musculoskeletal Diseases; Mental Disorder
MeSH Terms: conditions — Musculoskeletal Diseases; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Sick-listed employees with musculoskeletal disorders and/or common mental disorders will receive an invitation to the study from the labor-and welfare administration. Individuals who consent to participate will be allocated to either treatment as usual or personalized advice from an expert-team.
Who Masked: Outcomes Assessor
Masking Description: It is not possible to blind the participants or the care providers. As the investigators also will be care providers in this study, they will also have knowledge of the allocation.
  After the intervention, all data will be depersonalized and the name and other identifiers will be replaced by a study number. The outcome will be collected from national registries and the merging of data will be done by a statistician in the labor- and welfare administration who is not involved in the assessment of data. This allows the researchers to be blinded when they analyze the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital expert team (Experimental): The participants allocated to this arm will receive personalized advice from an expert team. The participants will have one video meeting with the team and receive a written report.
  Interventions: Procedure: Digital expert team
- Treatment as usual (No Intervention): The participants will answer a digital questionnaire and will get normal follow-up from his/her general practitioner and labor- and welfare administration (NAV).

INTERVENTIONS:
Procedure: Digital expert team — A digital team will be appointed based on the participant's answers in the digital screening questionnaire. Members of the team can be specialists in Physical and rehabilitation medicine, psychologist, physiotherapist, social workers, and consultants in the labor- and welfare administration. The general practitioner will also be invited to the meeting.
  Arms: Digital expert team

SUMMARY:
Long-term sick leave is a challenge in Norway, and the healthcare and labor- and welfare services are often not coordinated in helping the sick-listed employees return to work. In this study, the investigators want to evaluate the effectiveness of an intervention where an expert team provides advice for an individualized patient pathway based on information from a digital questionnaire and a video meeting with the sick-listed employee and the participant's general practitioner. The patient pathway should include both healthcare and labor- and welfare services measures.

Sick-listed patients with musculoskeletal- and/or common mental disorders are invited to join the study. They will receive a digital questionnaire and be randomized to either treatment as usual or personalized advice from an expert team. The team will be put together based on the response from the individual's questionnaire.

The investigators will evaluate the effect on return to work and the use of health care services 12 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Sick-listed minimum 50% between 11 and 20 weeks
* Musculoskeletal disorder and/or common mental disorder
* Living in the county of Trøndelag or Møre- og Romsdal

Exclusion Criteria:

* Specific conditions such as fracture, trauma, infections, malignancy, dislocations, etc.
* Serious mental conditions or another serious disease that makes participation difficult
* Most likely to return to work within 2 weeks
* Not speaking/reading Norwegian

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Return to work | 12 months
  Time to return to work within 12 months for at least 4 consecutive weeks

SECONDARY OUTCOMES:
Function | 12 months
  Approvement in function measured by Versus Arthritis Musculoskeletal Health Questionnaire (MSK-HQ). The MSK-HQ is scored on a range of 0-56, with a better score indicating better MSK-HQ health status
Change in pain | 12 months
  Change in pain measured on a numeric rating scale (0-10), with a higher score indicating more pain
Change in depression symptoms | 12 months
  Improvement in depression symptoms measured by Patient Health Questionnaire-9 (PHQ-9). PHQ-9 is scored on a range of 0-27, with higher score indicating more serious symptoms
Change in anxiety symptoms | 12 months
  Improvement in anxiety symptoms measured by Generalized Anxiety Disorder 7-item (GAD-7). GAD-7 is scored on a range of 0-21, with higher score indicating more serious symptoms
Days lost from work | 12 months
  Lost workdays during one year after intervention

OTHER OUTCOMES:
Sleep quality and insomnia | 12 months
  Prevalence of insomnia and bad sleep quality and change after 12 months. Measured with Insomnia severity index (ISI). ISI is scored on a range from 0-4, with higher score indicating more serious symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Gunn Hege Marchand, PhD, Study Director — St. Olavs hospital HF
Locations (4):
- Norway (4):
  - Ålesund sjukehus, Ålesund, Midt-Norge
  - Sykehuset Levanger, Levanger, Midt-Norge
  - Molde Sjukehus, Molde, Midt-Norge
  - St. Olavs hospital HF, Trondheim, Midt-Norge

IPD SHARING:
Plan to Share IPD: No